CLINICAL TRIAL: NCT06373549
Title: Investigation of the Protective Effects of Cardioplegia Solutions Used in Open Heart Surgery on Myocardial Redox Homeostasis at the Level of Redox System and Antioxidant System
Brief Title: Investigation of Myocardial Protection Efficacy of Cardioplegia Solutions Used in Open Heart Surgery
Status: Completed | Type: Observational
Sponsor: Tamer cebe (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Tamer cebe, Asistant Doctor, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Organization: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Other Study IDs: 2022/183-3896
Record Dates: First submitted 2024-02-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Myocardial Reperfusion Injury
Keywords: cardioplegia; del Nido; open heart surgery; oxidative stress; redox status
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with coronary artery bypass surgery due to coronary artery disease: From the patients included in the study, blood samples will be taken from the systemic venous circulation before the operation, and from the coronary sinus at 4 minutes before and after the cross-clamp, via a retrograde cardioplegia cannula into yellow capped gel tubes.
  Interventions: Procedure: Patients with coronary artery bypass surgery routine procedural administration of cardioplegia solutions; Procedure: Patients who underwent heart valve surgery without coronary artery disease routine procedural administration of cardioplegia solutions
- Patients who underwent heart valve surgery without coronary artery disease: From the patients included in the study, blood samples will be taken from the systemic venous circulation before the operation, and from the coronary sinus at 4 minutes before and after the cross-clamp, via a retrograde cardioplegia cannula into yellow capped gel tubes.
  Interventions: Procedure: Patients with coronary artery bypass surgery routine procedural administration of cardioplegia solutions; Procedure: Patients who underwent heart valve surgery without coronary artery disease routine procedural administration of cardioplegia solutions

INTERVENTIONS:
Procedure: Patients with coronary artery bypass surgery routine procedural administration of cardioplegia solutions — To investigate the effectiveness of myocardial protection methods, blood samples were collected from the coronary sinus before the aortic cross-clamping and at 4 minutes after aortic cross-clamping, through a coronary sinus cannula with a yellow-capped gel tube. The collected blood samples were kept in an upright position for 20 minutes to allow separation into serum fraction, then centrifuged at 3000 g for 10 minutes (Beckman Coulter, Microfuge 16, USA). The obtained serums were aliquoted into 250 μl portions in Eppendorf tubes, separately for each patient.
Procedure: Patients who underwent heart valve surgery without coronary artery disease routine procedural administration of cardioplegia solutions — To investigate the effectiveness of myocardial protection methods, blood samples were collected from the coronary sinus before the aortic cross-clamping and at 4 minutes after aortic cross-clamping, through a coronary sinus cannula with a yellow-capped gel tube. The collected blood samples were kept in an upright position for 20 minutes to allow separation into serum fraction, then centrifuged at 3000 g for 10 minutes (Beckman Coulter, Microfuge 16, USA). The obtained serums were aliquoted into 250 μl portions in Eppendorf tubes, separately for each patient.

SUMMARY:
Cardioplegias are different pharmacokinetic solutions routinely used in cardiac surgery to protect the heart from ischemia and induce arrest. Various cardioplegia solutions (such as Bretschneider, del Nido, blood cardioplegia, crystalloid cardioplegia, St. Thomas) are used in clinical practice. There is no clear scientific data in the literature that demonstrates the superiority of one cardioplegia over the others. The choice of the appropriate cardioplegia depends on the surgeon's clinical experience and preference. In this study preferred the blood cardioplegia and del Nido cardioplegia, which are commonly used in clinic. Both cardioplegias have different advantages that contribute to their preference in clinical practice.

Blood cardioplegia is an autologous cardioplegia that includes physiological buffer systems, allowing for heart nourishment and containing native antioxidant systems. However, the need for repeated doses every 20 minutes after the initial application creates a disadvantage in terms of surgical comfort. On the other hand, del Nido cardioplegia is preferred by surgeons in complex cases due to its long application intervals. The adequacy of a single dose for up to 90 minutes after the initial application creates an advantage in terms of surgical comfort and surgical integrity. However, the content being predominantly electrolyte-based, containing 1:4 ratio of autologous blood, and the extended time of a single dose are disadvantages compared to blood cardioplegia in terms of heart nourishment and protection from ischemia. In addition to these different usage scenarios, the myocardial protective effects of cardioplegias on cellular redox homeostasis are also among the current research topics. Thesis project can contribute to the current literature and clinical practice on the cardioprotective advantages of cardioplegia solutions and the reasons for their preference in surgery.

DETAILED DESCRIPTION:
Cardioplegias are routinely used in cardiac surgery to protect the heart from ischemia. Choice of the cardioplegia depends on surgeons clinical experience and preference. Various cardioplegia solutions (such as Bretschneider, del Nido, blood cardioplegia, crystalloid cardioplegia, St. Thomas) are widely used in clinical practice. There is no clear scientific data in the current literature that demonstrates the superiority of one cardioplegia over the others.

In this study preferred the blood and del Nido cardioplegia solutions, which are commonly used in clinic. Blood cardioplegia is an autologous cardioplegia that includes physiological buffer systems, allowing for heart nourishment and containing native antioxidant systems. However, the need for repeated doses every 20 minutes after the initial application creates a disadvantage in terms of surgical comfort. On the other hand, del Nido cardioplegia is preferred by surgeons in complex cases due to its long application intervals.

The adequacy of a single dose for up to 90 minutes after the initial application creates an advantage in terms of surgical comfort and surgical integrity. However, the content being predominantly electrolyte-based, containing 1:4 ratio of autologous blood, and the extended time of a single dose are disadvantages compared to blood cardioplegia in terms of heart nourishment and protection from ischemia. Hamad et al reported that del Nido and blood cardioplegia solutions offer equivalent safety in combined adult valve surgery. In addition to these differences, the myocardial protective effects of cardioplegias on myocardial redox homeostasis are also among the current research topics. Ischemia and reperfusion injury can be observed in the myocardial tissues of patients undergoing coronary artery bypass graft surgery and isolated valve replacement surgery. It was reported that coronary sinus blood sampling gives an insight into the localized pathophysiology of heart diseases. Comparative research examining the effects of blood and del Nido cardioplegia solutions on coronary sinus redox status is not currently available in the literature. The study aim to contribute to the development of effective strategies to minimize oxidative damage associated with cardiac surgery by investigating the effects of blood and del Nido cardioplegia solutions on coronary sinus redox homeostasis during the preoperative and postoperative periods using redox biomarkers and antioxidant system transcription factors. Thesis project also intend to compare these redox effects with elective isolated valve replacement surgery patients, who do not have coronary artery disease but share a similar pathogenesis with potential strategies for minimizing oxidative damage associated with cardiac surgery using cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective coronary artery bypass surgery due to coronary artery disease
* Patients without coronary artery disease who underwent elective valve surgery
* Patients between the ages of 18-75
* Having a BMI of 18.5-30

Exclusion Criteria:

* Being under 18 years old
* Patients older than 75 years
* Patients requiring valve surgery (combined surgical procedure) with coronary artery bypass
* Patients who underwent emergency coronary bypass
* BMI > 30 obese patients

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital, Adult Cardiovascular Surgery Clinic will be selected among the patients who will undergo cardiac surgery and meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Evaluation of the myocardial protective effects of different cardioplegia solutions through oxidative stress and redox signaling molecules. | 1-7 days
  The PCO concentration was expressed as nmol/mg protein. The standard curve was used to express the AOPP concentrations as micromoles per liter of chloramine-T equivalents.Lipid peroxidation rate of coronary sinus blood samples was assessed with a calibration curve for peroxide value using xylenol orange and Fe3+ chloride.
  Mitochondrial superoxide dismutase expression.MnSOD concentrations of the coronary sinus blood samples were expressed as ng/mL.GPx activities of the coronary sinus blood samples were expressed as U/mg protein.The CAT activity is measured as the difference in absorbance per unit time.CAT concentrations of the coronary sinus blood samples were expressed as KU/L.The serum Nrf2 levels of the samples were expressed as ng/L.The serum Keap1 levels of the samples were expressed as ng/L.The samples' serum PGC-1α levels were reported as ng/mL.

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ. Dr. Siyami Ersek Göğüs Kalp ve Damar Cerrahisi Eğitim ve Araştırma Hastanesi Erişkin Kalp ve Damar Cerrahisi Kliniği, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
During the process of obtaining informed consent from the participants involved in the study, it was stated that their data would not be used elsewhere.

REFERENCES:
- [Background] Carvajal C, Goyal A, Tadi P. Cardioplegia. 2023 Jul 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554463/ PMID 32119350
- [Background] Comentale G, Giordano R, Palma G. Comparison of the different cardioplegic strategies in cardiac valves surgery: who wins the "arm-wrestling"? J Thorac Dis. 2018 Feb;10(2):714-717. doi: 10.21037/jtd.2018.01.133. No abstract available. PMID 29607140
- [Background] Weber C, Jenke A, Chobanova V, Yazdanyar M, Chekhoeva A, Eghbalzadeh K, Lichtenberg A, Wahlers T, Akhyari P, Paunel-Gorgulu A. Targeting of cell-free DNA by DNase I diminishes endothelial dysfunction and inflammation in a rat model of cardiopulmonary bypass. Sci Rep. 2019 Dec 17;9(1):19249. doi: 10.1038/s41598-019-55863-8. PMID 31848423
- [Background] Atayik MC, Cakatay U. Redox signaling and modulation in ageing. Biogerontology. 2023 Oct;24(5):603-608. doi: 10.1007/s10522-023-10055-w. Epub 2023 Aug 3. PMID 37535201
- [Background] Ulasov AV, Rosenkranz AA, Georgiev GP, Sobolev AS. Nrf2/Keap1/ARE signaling: Towards specific regulation. Life Sci. 2022 Feb 15;291:120111. doi: 10.1016/j.lfs.2021.120111. Epub 2021 Oct 31. PMID 34732330
- [Background] Calabrese EJ, Kozumbo WJ. The hormetic dose-response mechanism: Nrf2 activation. Pharmacol Res. 2021 May;167:105526. doi: 10.1016/j.phrs.2021.105526. Epub 2021 Mar 2. PMID 33667690
- [Background] GIBBON JH Jr. Application of a mechanical heart and lung apparatus to cardiac surgery. Minn Med. 1954 Mar;37(3):171-85; passim. No abstract available. PMID 13154149
- [Background] Topcu AC, Bolukcu A, Ozeren K, Kavasoglu T, Kayacioglu I. Normoxic management of cardiopulmonary bypass reduces myocardial oxidative stress in adult patients undergoing coronary artery bypass graft surgery. Perfusion. 2021 Apr;36(3):261-268. doi: 10.1177/0267659120946733. Epub 2020 Aug 5. PMID 32755372
- [Background] Cebe T, Yanar K, Atukeren P, Ozan T, Kuruc AI, Kunbaz A, Sitar ME, Mengi M, Aydin MS, Esrefoglu M, Aydin S, Cakatay U. A comprehensive study of myocardial redox homeostasis in naturally and mimetically aged rats. Age (Dordr). 2014;36(6):9728. doi: 10.1007/s11357-014-9728-y. Epub 2014 Nov 11. PMID 25384832
- [Background] Cebe T, Atukeren P, Yanar K, Kuruc AI, Ozan T, Kunbaz A, Sitar ME, Mirmaroufizibandeh R, Aydin S, Cakatay U. Oxidation scrutiny in persuaded aging and chronological aging at systemic redox homeostasis level. Exp Gerontol. 2014 Sep;57:132-40. doi: 10.1016/j.exger.2014.05.017. Epub 2014 May 28. PMID 24879971